CLINICAL TRIAL: NCT01283217
Title: A Randomized, Multicenter, Open-label, Phase III Trial of Docetaxel and S1 (DS) Versus S1 and Cisplatin (SP) in Curatively Resected (D2) Gastric Cancer of Stage IIIB/IV (M0)
Brief Title: Docetaxel and S1 (DS) Versus S1 and Cisplatin (SP) in Curatively Resected Stage IIIB/IV Gastric Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 4-2009-0708
Record Dates: First submitted 2011-01-24; First posted 2011-01-25 (Estimated); Last update posted 2013-06-04 (Estimated); Status verified 2013-06

CONDITIONS: Gastric Adenocarcinoma
MeSH Terms: interventions — S 1 (combination); Docetaxel; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DS(Docetaxel with S-1) (Experimental): Docetaxel with S-1
  Interventions: Drug: DS
- SP(S-1 with cisplatin) (Active Comparator): S-1 with cisplatin
  Interventions: Drug: SP

INTERVENTIONS:
Drug: DS — Docetaxel with S-1. S-1: Orally, within 30 minutes after ingestion of food. Docetaxel and Cisplatin: IV infusion.
  Other Names: Test group : DS * 8 cycles; (S-1 70mg/m2/D, D1~14 plus Docetaxel 35 mg/m2 D1,8 q 3weeks)
  Arms: DS(Docetaxel with S-1)
Drug: SP — S-1 with cisplatin. S-1 : Orally, within 30 minutes after ingestion of food. Docetaxel and Cisplatin: IV infusion.
  Other Names: Control group : SP * 8 cycles; (S-1 70mg/m2/D, D1~14 + Cisplatin 60mg2 D1, q 3 weeks)
  Arms: SP(S-1 with cisplatin)

SUMMARY:
Docetaxel was the first drug that showed survival benefits when added to the CF regimen, but it was very toxic. Docetaxel is also has a synergistic anti-cancer effect with S-1, in phase I/II studies. The use of a docetaxel plus S-1 combination as first-line chemotherapy for advanced gastric cancer achieved response rates of 46~56% and a median survival time of 14.0~14.3 months.

Based upon this background, the aim of this study is to detect a significant increase in 3 year DFS of disease for the test group (DS) relative to the Control group (SP).

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven, Stage IIIb/ IIIc curatively resected gastric carcinoma
* ECOG performance status 0-1
* Curatively resected advanced gastric cancer patients of stage IIIb/IIIc
* D2 lymph node dissection with R0 surgery
* Signed informed consent

Exclusion Criteria:

* Subjects with documented distant metastasis.
* Malabsorption syndrome or disease significantly affecting gastrointestinal function
* Patients with other uncontrolled systemic illness, e.g. infection, poorly controlled HTN
* History of other malignancy. Subjects who have been disease-free for 5 years or subjects with successfully treated in situ carcinoma are eligible.
* Subjects with preoperative/adjuvant other cancer treatment, such as chemotherapy, immunotherapy and radiotherapy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Estimated)
Dates: Start 2010-03; Primary Completion 2016-03 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
3-year disease free survival(DFS) | 3 years
  Tumor assessments with chest X-rays and CT or MRI scan will be done at 6 months after randomization (after the end of the treatment period), then every 3 months for the first 2 years after randomization and then every 6 months for coming 3 years then one year basis until completion of the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, South Korea